CLINICAL TRIAL: NCT03708614
Title: A Feasibility and Acceptability Study of Elevated Protein Dietary Intake for Children Diagnosed With Autism Spectrum Disorder (ASD) While on Atypical Antipsychotic Medication
Brief Title: A Study Looking at How Well Children With Autism Spectrum Disorder on Medications Like Having More Protein
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Lorry Chen, Clinical Dietitian, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB 18-781
Record Dates: First submitted 2018-10-02; First posted 2018-10-17 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Atypical antipsychotic medication; Psychotropic medication; Psychotropic-induced weight gain; Controlled energy intake with elevated protein; Dietary intervention; Acceptability; Feasibility
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Non-randomized pilot intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled energy intake with elevated protein intake (Other): Dietary intervention - Participants will be counseled to elevate protein and control energy intake for ten consecutive weeks.
  Interventions: Other: Controlled energy diet with elevated protein intake

INTERVENTIONS:
Other: Controlled energy diet with elevated protein intake — Participants will be counseled to elevate protein and control energy intake for ten consecutive weeks. Protein intake will be increased in the range of 20-30% of total daily caloric intake. Each participant's diet will also be modified to implement controlled energy intake. Controlled energy intake will be defined as being isocaloric with the participant's current dietary intake.

SUMMARY:
Antipsychotic medications are commonly prescribed in children and adults with ASD (Curtin, Jojic & Bandini, 2014). But weight gain has been known to be one of the less desirable effects of these medications, increasing one's risk for overweight and obesity. Based on experience in Holland Bloorview's Nutrition Clinic, working with a dietitian to follow specific dietary advice, such as having more protein while keeping the amount of calories the same, may be a possible and useful way to limit weight gain.

This study's objective is to evaluate the feasibility (study designs, methods, processes) and acceptability (client/family satisfaction, perceived effectiveness) of a controlled energy diet with elevated protein intake in children and youth with ASD who are currently taking prescribed atypical antipsychotic medication.

DETAILED DESCRIPTION:
The use of psychotropic medication in children and youth with Autism Spectrum Disorder (ASD) to treat symptoms of aggression, irritability and related behavioural problems has become increasingly common in recent years. Data obtained from clinical and nationally representative populations of children demonstrate that approximately 30%-60% of children with ASD are prescribed at least one psychotropic medication, and 10% are prescribed more than three medications at the same time (Curtin, Jojic & Bandini, 2014).

Weight gain, which is one of the harmful effects of psychotropic medication, is likely one of the most understood risk factors for obesity in children and adults with ASD. In a systematic review and meta-analysis of double-blinded, randomized, controlled trials studying the metabolic adverse effects of atypical antipsychotics in children and adolescents under 18 years of age, risperidone, olanzapine and aripiprazole were associated with statistically significant weight gain compared with placebo (Almandil et al., 2013). Similar findings were reported from a review of literature, using PubMed, on weight gain and increase of BMI among children and adolescents (0-18 years old) treated with antipsychotic medications (Martinez-Ortega et al., 2013).

Although clinical trials with different agents have been conducted in an attempt to address weight gain in individuals on psychotropic medications, no established treatments or preventative measures have been developed to combat psychotropic-induced weight gain (PIWG) to date (Curtin, Jojic & Bandini, 2014). A review of published literature using PubMed yielded limited and mixed results for using Metformin as the intervention for the treatment in combating PIWG (Anagostou et al., 2016; Handen et al., 2017). Based on clinical experience in Holland Bloorview's Nutrition Clinic, controlled energy intake combined with elevated protein intake (CEEP) may represent an effective and practical strategy for limiting weight gain.

Potential beneficial outcomes associated with protein ingestion include: a) increased satiety, which is being satisfactorily full - protein generally increases satiety to a greater extent than carbohydrate or fat and may facilitate a reduction in energy consumption; b) increased thermogenesis, which is the production of heat in the body - higher protein diets are associated with an increase in thermogenesis, which also influences satiety and increases energy expenditure; and c) maintenance or growth of fat-free mass (muscle) - an elevated protein diet may provide an increase effect on muscle protein synthesis in some individuals, favouring the retention of lean muscle mass while improving metabolic profile (Paddon-Jones et al., 2018).

This study's primary objective is to evaluate the feasibility (study designs, methods, processes) and acceptability (client/family satisfaction, perceived effectiveness) of a controlled energy diet with elevated protein intake in children and youth with ASD who are currently taking prescribed atypical antipsychotic medication.

Children and youth, ages 6-17 years old, with ASD (n=10) on atypical antipsychotic medication will be exposed to specific nutrition recommendations involving CEEP for ten consecutive weeks. Each participant and parent/guardian will work collaboratively with the RD/RA to formulate strategies to slowly increase protein intake in the range of 20-30% of total caloric intake and ensure consistent energy intake. Data will be collected through food records, anthropometric measurements and informal post-intervention interviews to measure the feasibility and acceptability of the study processes and elevated protein dietary changes.

ELIGIBILITY:
Inclusion Criteria:

1. Child Inclusion Criteria:

   * Diagnosis of ASD
   * Currently taking one or more atypical antipsychotic medication
   * Ages 6-17 years old
   * Enrolment as an active client in a Psychopharmacology Clinic at Holland Bloorview
   * Accepts all food, based on the SOS Feeding Approach: Defining Picky vs. Problem Eaters by Kay Toomey (2017) - has no significant food aversions; will accept new foods on plate, usually can touch or taste; and consumes one or more foods from all food groups, varying in textures
   * Can communicate in English
   * Has access to a telephone
2. Parent/guardian inclusion criteria:

   * Provides care to study participant
   * Can communicate in English
   * Able to complete food records
   * Has access to a telephone

Exclusion Criteria:

a) Child exclusion criteria:

* Medical condition that contradicts elevated protein intake
* Has significant food aversions
* Has any food allergies
* Currently participating in another clinical study that would interfere with anticipated endpoints and outcome measurements

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Caloric and protein intake | At the time of study enrolment (week 0) and during week 10 of intervention implementation (week 10)
  Average caloric (kcal) and protein (g) intake - comparison of three day food records measured at the time of enrolment and during week 10 of intervention implementation
Pre- (at time of study enrolment) and post-intervention anthropometric measurements | Measured at the time of study enrolment (week 0) and after ten weeks of intervention (week 11), assessed up to 11 weeks
  Weight in kilograms - to calculate weight changes and BMI
Pre- (at time of study enrolment) and post-intervention anthropometric measurements | Measured at the time of study enrolment (week 0) and after ten weeks of intervention (week 11), assessed up to 11 weeks
  Height in centimetres - to calculate BMI
Pre- (at time of study enrolment) and post-intervention anthropometric measurements | Measured at the time of study enrolment (week 0) and after ten weeks of following the intervention (week 11), assessed up to 11 weeks
  Skinfold (triceps and subscapular) measurements in millimetres
Post-intervention interview with participants and family | Interview (anticipated duration of 60 minutes) will be conducted after week ten of intervention implementation (week 11)
  Qualitative interview (guided using semi-structured format) to gain insight into successful strategies and potential barriers to consistently implement elevated protein dietary changes
Study feasibility (designs, methods, processes) | During the screening and recruitment process (anticipated duration of 1-1.5 months)
  Recruitment rates - comparisons between (i) number of patients screened; (ii) number of eligible patients identified from clinic; (iii) number of eligible patients approached; (iv) number of patients who agreed to further contact; and (v) number of participants consented and enrolled in the study.
Study feasibility (designs, methods, processes) | Measurements taken at the start of the study during enrolment and at study completion (anticipated duration of 5 months)
  Retention rate - comparison between (i) number of participants enrolled at the start of the study; and (ii) number of participants enrolled at the end of study.
Study feasibility (designs, methods, processes) | Measured at the time of study enrolment (week 0) and after ten weeks of intervention (week 11), assessed up to 11 weeks
  Completion rates - Number of participants who completed the three-day food records
Study feasibility (designs, methods, processes) | Interview (anticipated duration of 60 minutes) will be conducted after week ten of intervention implementation (week 11)
  Qualitative interview (guided using semi-structured format) to assess the participants' perspectives on the acceptability and feasibility of completing food records
Study feasibility (designs, methods, processes) | Interview (anticipated duration of 60 minutes) will be conducted after week ten of intervention implementation (week 11)
  Qualitative interview (guided using semi-structured format) to assess the participants' perspectives on the acceptability and feasibility of attending on-site visits for anthropometric measurements
Study feasibility (designs, methods, processes) | Interview (anticipated duration of 60 minutes) will be conducted after week ten of intervention implementation (week 11)
  Qualitative interview (guided using semi-structured format) to assess the participants' perspectives on the acceptability and feasibility of following-up with the RA via phone during intervention implementation
Study feasibility (designs, methods, processes) | Interview (anticipated duration of 60 minutes) will be conducted after week ten of intervention implementation (week 11)
  Qualitative interview (guided using semi-structured format) to assess the participants' perspectives on the acceptability and feasibility of participating in the on-site post-intervention interview

CONTACTS AND LOCATIONS:
Overall Officials: Lorry Chen, Honors BSc., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as all study data will be de-identified and coded after the recruitment process. Only members of the research team will have access to the research data and linking log. The key-code will be deleted at the end of the study. Results from the study will be disseminated through publication, written lay summary and knowledge translation communication products.

REFERENCES:
- [Background] Almandil NB, Liu Y, Murray ML, Besag FM, Aitchison KJ, Wong IC. Weight gain and other metabolic adverse effects associated with atypical antipsychotic treatment of children and adolescents: a systematic review and meta-analysis. Paediatr Drugs. 2013 Apr;15(2):139-50. doi: 10.1007/s40272-013-0016-6. PMID 23519708
- [Background] Anagnostou E, Aman MG, Handen BL, Sanders KB, Shui A, Hollway JA, Brian J, Arnold LE, Capano L, Hellings JA, Butter E, Mankad D, Tumuluru R, Kettel J, Newsom CR, Hadjiyannakis S, Peleg N, Odrobina D, McAuliffe-Bellin S, Zakroysky P, Marler S, Wagner A, Wong T, Macklin EA, Veenstra-VanderWeele J. Metformin for Treatment of Overweight Induced by Atypical Antipsychotic Medication in Young People With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2016 Sep 1;73(9):928-37. doi: 10.1001/jamapsychiatry.2016.1232. PMID 27556593
- [Background] Curtin C, Jojic M, Bandini LG. Obesity in children with autism spectrum disorder. Harv Rev Psychiatry. 2014 Mar-Apr;22(2):93-103. doi: 10.1097/HRP.0000000000000031. PMID 24614764
- [Background] Handen BL, Anagnostou E, Aman MG, Sanders KB, Chan J, Hollway JA, Brian J, Arnold LE, Capano L, Williams C, Hellings JA, Butter E, Mankad D, Tumuluru R, Kettel J, Newsom CR, Peleg N, Odrobina D, McAuliffe-Bellin S, Marler S, Wong T, Wagner A, Hadjiyannakis S, Macklin EA, Veenstra-VanderWeele J. A Randomized, Placebo-Controlled Trial of Metformin for the Treatment of Overweight Induced by Antipsychotic Medication in Young People With Autism Spectrum Disorder: Open-Label Extension. J Am Acad Child Adolesc Psychiatry. 2017 Oct;56(10):849-856.e6. doi: 10.1016/j.jaac.2017.07.790. Epub 2017 Aug 19. PMID 28942807
- [Background] Martinez-Ortega JM, Funes-Godoy S, Diaz-Atienza F, Gutierrez-Rojas L, Perez-Costillas L, Gurpegui M. Weight gain and increase of body mass index among children and adolescents treated with antipsychotics: a critical review. Eur Child Adolesc Psychiatry. 2013 Aug;22(8):457-79. doi: 10.1007/s00787-013-0399-5. Epub 2013 Mar 17. PMID 23503976
- [Background] Paddon-Jones D, Westman E, Mattes RD, Wolfe RR, Astrup A, Westerterp-Plantenga M. Protein, weight management, and satiety. Am J Clin Nutr. 2008 May;87(5):1558S-1561S. doi: 10.1093/ajcn/87.5.1558S. PMID 18469287